CLINICAL TRIAL: NCT01667432
Title: A Multicenter, Prospective, Observational, Non-interventional Study Evaluating On-treatment Predictors of Response in Subjects With HBeAg Positive or HBeAg Negative Chronic Hepatitis B Receiving Therapy With PEGASYS® (Peginterferon Alfa-2a 40KD)
Brief Title: An Observational Study of Peginterferon Alfa-2a (PEGASYS®) in Patients With HBeAg Positive or HBeAg Negative Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25626
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Peginterferon alfa-2a: Participants received peginterferon alfa-2a (PEGASYS®) 180 µg subcutaneously in the abdomen or thigh once weekly for 12 weeks.
  Interventions: Biological: Peginterferon alfa-2a

INTERVENTIONS:
Biological: Peginterferon alfa-2a — Peginterferon alfa-2a commercial product (PEGASYS®) was supplied as a solution in prefilled syringes.
  Other Names: PEGASYS®; RO0258310

SUMMARY:
This prospective, multicenter, observational study will evaluate on-treatment predictors of response in patients with HBeAg positive or HBeAg negative chronic hepatitis B receiving treatment with peginterferon alfa-2a (PEGASYS®) in accordance with local labeling and the summary of product characteristics. Data will be collected from patients for the duration of their treatment and for up to 24 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age.
* Hepatitis B envelope antigen (HBeAg) positive or HBeAg negative hepatitis B with or without cirrhosis.
* Elevated alanine aminotransferase (ALT) > upper limit of normal (ULN) but ≤ 10 x ULN according to local label.

Exclusion Criteria:

* Contraindications to peginterferon alfa-2a (PEGASYS®) as detailed in the label.
* Co-infection with hepatitis A, hepatitis C, or human immunodeficiency virus (HIV).
* Concomitant treatment with telbivudine.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B on treatment with PEGASYS.
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2011-07-08 (Actual); Primary Completion 2014-08-12 (Actual); Study Completion 2014-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Bulgaria (9):
  - Mhat - Pleven; Clinic of Gastroenterology, Pleven
  - Umhat St. Georgi; Clinical of Gastroenterology, Plovdiv
  - MHAT Tokuda Hospital Sofia; Department of Gastroenterology at Clinic of Internal Deseases, Sofia
  - UMHAT Alexandrovska EAD; Gastroenterology, Sofia
  - Mhat Queenjoanna; Clinic of Gastroenterology, Sofia
  - Military Medical Academy; Gastroenterology, Sofia
  - Mhat St. Ivan Rilski; Clinic of Gastroenterology, Sofia
  - Mhat St. Zagora; Clinical of Gastroenterology, Stara Zagora
  - Mhat Sveta Marina; Clinic of Gastroenterology, Varna

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a
Started | 141
Completed | 84
Not Completed | 57
Not completed — Premature Study Termination | 26
Not completed — Failure to Return | 10
Not completed — Moved to Another Center | 3
Not completed — Lost to Follow-up | 3
Not completed — Refused Treatment/Withdrew Consent | 1
Not completed — Insufficient Therapeutic Response | 4
Not completed — Adverse Event | 1
Not completed — Protocol Deviation | 2
Not completed — Principal Investigator Decision | 1
Not completed — Reason Not Specified | 2
Not completed — Missing Information | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All participants who received at least 1 dose of peginterferon alfa-2a.
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.10 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 119

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Suppression of HBV DNA to < 2,000 IU/ml at the End of the Study
Description: Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) was assessed in plasma samples using quantitative polymerase chain reaction (PCR). Results are reported in international units (IU) per milliliter (ml).
Time Frame: At the end of the study (Week 36)
Population: Intent-to-treat population: All participants who received at least 1 dose of peginterferon alfa-2a.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Peginterferon Alfa-2a: Intent-to-treat population: All participants who received at least 1 dose of peginterferon alfa-2a.
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 139
Percentage of participants | 38.8 [30.70 to 47.48]

2. Primary Outcome: Percentage of Patients With Suppression of HBV DNA < 2,000 IU/ml
Time Frame: approximately 3 years
Reporting Status: Not Posted

3. Secondary Outcome: Percentage of Participants With Suppression of HBV DNA to < 80 IU/ml at the End of Treatment
Description: Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) was assessed in plasma samples using quantitative polymerase chain reaction (PCR). Results are reported in international units (IU) per milliliter (ml) separately for participants who were hepatitis B envelope antigen (HBeAg) positive and HBeAg negative.
Time Frame: At the end of treatment (Week 24)
Population: Intent-to-treat population: All participants who received at least 1 dose of peginterferon alfa-2a. Only participants with available HBsAg measurements were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 37
percentage of participants
  HBeAg positive (n = 4) | 36.4 [10.92 to 69.21]
  HBeAg negative (n = 33) | 26.6 [19.8 to 35.3]

4. Secondary Outcome: HBsAg Clearance: Percentage of Patients Who Become HBsAg Negative
Time Frame: approximately 3 years
Reporting Status: Not Posted

5. Secondary Outcome: Correlation of HBsAg Clearance With Other On-treatment Factors in HBeAg Positive and HBeAg Negative Patients
Time Frame: approximately 3 years
Reporting Status: Not Posted

6. Secondary Outcome: Correlation of HBsAg Clearance With Pre-treatment Factors in HBeAg Positive and HBeAg Negative Patients
Time Frame: approximately 3 years
Reporting Status: Not Posted

7. Secondary Outcome: Incidence of Serum ALT Normalization: Serum ALT/ALT Ratio
Time Frame: approximately 3 years
Reporting Status: Not Posted

8. Primary Outcome: In HBeAg Positive Patients: Percentage of Patients Who Become HBeAg Negative and Anti-HBe Positive
Time Frame: approximately 3 years
Reporting Status: Not Posted

9. Secondary Outcome: Safety: Incidence of Adverse Events
Time Frame: approximately 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safety population: All participants who received at least 1 dose of peginterferon alfa-2a and had at least 1 post-baseline safety assessment.
Arm/Group | Peginterferon Alfa-2a
Serious Adverse Events (participants affected / at risk) | 1/139
Other Adverse Events (participants affected / at risk) | 78/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alfa-2a (N=139)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alfa-2a (N=139)
Fever (General disorders) | 42 (42)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (27)
Leucopenia (Blood and lymphatic system disorders) | 23 (23)
Hypertransaminasaemia (Hepatobiliary disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.